CLINICAL TRIAL: NCT07160491
Title: Early Pre-hospital Thrombolysis Guided by Artificial Intelligence Assisted Mobile Application in Patients With ST-elevation Myocardial Infarction: A Multi-center Cluster Randomized Controlled Trial
Brief Title: Early Thrombolysis Guided by AI-Assisted App in Patients With STEMI
Acronym: EARLY-OPEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, MD, PhD, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EARLY-OPEN
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: Thrombolysis; appliaction; myocardial infarction; cluster randomized trial
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Multi-center, cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive promotion group (Experimental): A novel artificial intelligence assisted mobile application will be used in the experimental group to guide entire reperfusion process in patients with STEMI. The functions of the application include patient screening, education and training, route planning for patient transfer, time management, and quality control, etc.
  Interventions: Other: A novel artificial intelligence assisted mobile application
- Control group (No Intervention): Patients in the control group will be tranferred and managed according to the existing model

INTERVENTIONS:
Other: A novel artificial intelligence assisted mobile application — A novel artificial intelligence assisted mobile application will be used in the experimental group to guide entire reperfusion process in patients with STEMI. The functions of the application include patient screening, education and training, route planning for patient transfer, time management, and quality control, etc.The thrombolytic drug used in this study is tenecteplase (manufacturer: CSPC Pharmaceutical Group Limited, China ).
  Arms: Comprehensive promotion group

SUMMARY:
The aim of the study is to elucidate whether guiding by a novel artificial intelligence assisted mobile application can improve the clinical outcomes of patients in whom "guide wire passing through the lesion" could not be achieved within 120 min after diagnosis of STEMI, compared to conventional treatment strategies. With concerns of the inadequate use of thrombolysis in patients with STEMI in China, this study applies a new artificial intelligence assisted mobile application to guide the process of thrombolysis combined with PCI treatment, in order to accomplish the rapid coordination and cooperation of the whole medical network during re-perfusion treatment in different regions and different medical institutions in China, increases the proportion of early thrombolysis in pre-hospital setting, shortens the time from STEMI onset to reperfusion, and provides a reliable, effective and replicable new strategy for promoting and optimizing early reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* (the following inclusion conditions shall be met at the same time):

  1. age: ≥ 18 years and ≤ 80 years;
  2. Chest pain lasted for more than 30 min, and the onset time of chest pain was ≤ 12 hours;
  3. ECG: ST segment elevation after J-point in 2 or more adjacent leads: limb leads ≥ 0.1 mv or chest leads ≥ 0.2 mv;
  4. it is expected that "guide wire passing through the lesion" could not be achieved within 120 min after the diagnosis of STEMI;
  5. Signed informed consent .

Exclusion Criteria:

* (1) Cardiac rupture; (2) Complete left bundle branch block (LBBB) or ventricular pacing; (3) There are contraindications to thrombolysis; (4) Have serious comorbidities; (5) Have complex heart disease; (6) There are situations that are not suitable for clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3356 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse events (MAEs) at 1 year | Day 365
  Incidence of major adverse events (MAEs) at 1 year. MAE is a composite endpoint that includes all-cause mortality, stroke, cardiogenic shock, rehospitalization for ischemic heart failure, or reinfarction.

SECONDARY OUTCOMES:
Total ischemic time before reperfusion | Day 30
Total reperfusion rate during therapeutic time window | Hour 48
The proportion of ECG ST segment resolution（STR） ≥ 70% after thrombolysis or emergency PCI | Hour 48
Proportion of TIMI blood flow grade 3 before emergency PCI | Hour 48
Proportion of TIMI blood flow grade 3 after emergency PCI | Hour 48
Incidence of 30-day MAEs | Day 30
  MAE is a composite endpoint that includes all-cause mortality, stroke, cardiogenic shock, rehospitalization for ischemic heart failure, or reinfarction.
Incidence of major adverse cardiac events (MACE) at 1 year | Day 365
  MACE is a composite endpoint including cardiac death, reinfarction, clinically-driven revascularization, ischemic cardiomyopathy, or myocardial ischemia-driven rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD,PhD, Study Chair — Northern Theater Command General Hospital of the People's Liberation Army
Locations (1):
- No. 83, Wenhua Road, Shenhe District, Shenyang City, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No